CLINICAL TRIAL: NCT02562508
Title: Immunogenicity and Safety Study of a Bivalent Human Papillomavirus (Type 16, 18) Recombinant Vaccine (E.Coli) in Healthy Female Subjects Aged 9 to 17 Years
Brief Title: A Bridging Study of a Recombinant Human Papillomavirus 16/18 Bivalent Vaccine in Preadolescent Girls
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, professor, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPV-PRO-006
Record Dates: First submitted 2015-09-14; First posted 2015-09-29 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Vaginal Intraepithelial Neoplasia; Vulvar Intraepithelial Neoplasia; Persistent Infection
Keywords: Human Papilloma Virus 16; Human Papilloma Virus 18; vaccine; adolescent girl; bridging trial; non-inferiority
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 9-17y (0,1,6m) (Experimental): Participants in this arm would receive 60μg of HPV 16/18 bivalent vaccine according to 3 doses of HPV 16/18 bivalent vaccine
  Interventions: Procedure: 3 doses of HPV 16/18 bivalent vaccine
- 9-14y (0,6m) (Experimental): Participants in this arm would receive 60μg of HPV 16/18 bivalent vaccine according to 2 doses of HPV 16/18 bivalent vaccine
  Interventions: Procedure: 2 doses of HPV 16/18 bivalent vaccine
- 18-26y (0,1,6m) (Experimental): Participants in this arm would receive 60μg of HPV 16/18 bivalent vaccine according to 3 doses of HPV 16/18 bivalent vaccine
  Interventions: Procedure: 3 doses of HPV 16/18 bivalent vaccine

INTERVENTIONS:
Procedure: 3 doses of HPV 16/18 bivalent vaccine — Participants would receive 60μg of HPV 16/18 bivalent vaccine according to the standard 3-dose schedule (0,1,6 months)
  Arms: 18-26y (0,1,6m); 9-17y (0,1,6m)
Procedure: 2 doses of HPV 16/18 bivalent vaccine — Participants would receive 60μg of HPV 16/18 bivalent vaccine according to an alternative 2-dose schedule (0,6 months)
  Arms: 9-14y (0,6m)

SUMMARY:
This is a bridging trial of the recombinant HPV 16/18 bivalent vaccine manufactured by Xiamen Innovax Biotech CO., LTD.The primary objective of this study is to evaluate the immunogenicity (type specific IgG antibody) and safety of the tested vaccine administered in girls aged 9-17 years is non-inferior to young healthy adults of 18-26 years according to the standard 3-dose schedule (0,1,6 months). Meanwhile, this study tries to compare the difference of safety and immunogenicity among different schedules (0-6m vs 0-1-6m).

DETAILED DESCRIPTION:
Totally 750 healthy girls of 9-17 years and 225 healthy young women of 18-26 years were enrolled. The subjects of 9-14 years will be stratified into 2 subset. Subjects in each subsets will be randomly assigned into the standard 0-1-6m schedule group or an alternative 0-6m group. All subjects of 15-26 years of age will receive the standard 0-1-6m schedule. Participants were actively monitored for adverse events for 1 month after each injection. Severe adverse events during the trial were followed up. Serum samples from all the subjects would be collected on day 0, 6m, 7m to evaluate the immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged between 9 and 26 years when they receive the first vaccination (9≤age<27);
2. Participants aged 9-17 years whose legal guardian can provide identity certificate, or representative can provide authorization;
3. Judged as healthy and eligible for vaccination by the investigators through a self-reported medical history and some physical examinations;
4. Participants aged 9-17 years, able to sign or whose legal guardian agree to sign the written informed consent; or participants aged 18-26 years and agree to sign the written informed consent;
5. Able to comply with the requests of the study;
6. Axillary temperature not higher than 37.0°C;
7. Nonpregnancy verified by a urine pregnancy test;

Exclusion criteria:

1. Pregnant or lactating woman and any woman who are willing or intend to become pregnant in next 7 months;
2. Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first vaccination, or plan to use during the study period;
3. Participants who received an immunosuppressive agent or other immunomodulator agent for a long term (for 14 days or more) within 6 months of the first vaccination, or systematic corticosteroid (however, a topical corticosteroid is allowed, such as ointment, eye drops, inhalant, or nasal spray);
4. Participants who received immunoglobulin and/or blood product 3 months prior to the first vaccination, or planned to receive during the study period;
5. Use of any inactivated vaccine 14 days preceding dosing of study vaccine or attenuated vaccine 21 days before the enrollment;
6. Participants had fever (auxiliary temperature ≥38.0 °C) within 3 days prior to vaccination, or any acute disease requiring systematic antibiotics or antiviral therapy within the past 5 days;
7. Concurrently participating another clinical trial;
8. Participants who have received HPV vaccines;
9. Participants with immunodeficiency disease (such as HIV positive), primary disease in vital organs, cancer (or precancerous lesion), or chronic history of immunological disease requiring treatment (including systemic lupus erythematosus), rheumatoid arthritis, asplenia or splenectomy due to any conditions, and other immunological diseases that may impact immune response as considered by investigator), etc.;
10. Participants with a history of allergy, including severe adverse reactions due to the past vaccination, such as hypersensitivity, urticaria, dyspnea, angioneurotic edema, or abdominal pain;
11. Participants with asthma, which is unstable in the past 2 years, requiring emergency treatment, hospitalization, or oral or intravenous corticosteroid;
12. Participants with concurrent severe medical disorders, such as hypertension, heart disease, diabetes mellitus, or hyperthyroidism, etc.;
13. Participants with coagulation dysfunction (such as coagulation factor deficiency, blood-clotting disorder, or platelet disorder) or coagulation disorders, as diagnosed by a physician;
14. Participants with epilepsy, excluding febrile epilepsy in patients under 2 years old, alcoholic epilepsy 3 years prior to alcohol abstinence, or pure epilepsy requiring no treatment within the past 3 years;
15. Participants who are not compliant to the study's requirements due to psychological conditions, or those with prior or existing mental disease or bipolar psychosis which are not well controlled within the past 2 years and require taking drugs, or those with suicidal tendency within the past 5 years;
16. According to the investigator's judgment, there might be some medical, psychological, social or occupational factors which might impact on the individual to obey the protocol or sign the informed consent;

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 979 (Actual)
Dates: Start 2015-12-05 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2016-08-12 (Actual)

PRIMARY OUTCOMES:
Anti-HPV16 and anti-HPV18 seroconversion rates and geometric mean concentrations at Months 7 (type specific IgG antibody) | Month 7
  To detect the anti-HPV 16 and anti-HPV 18 type specific IgG antibody level on day 0 (before the 1st dose) ,six month after the dose 1 (before the 3rd dose) and one month after dose 3

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Month 7
  All the adverse events in one month after each dose would be recorded in the diary card. All the Serious Adverse Events(SAE) occurred during clinical trial time frame would be recorded.

OTHER OUTCOMES:
Anti-HPV16 and anti-HPV18 seroconversion rates and geometric mean concentrations at Months 7 (type specific neutralizing antibody) | Month 7
  To detect the anti-HPV 16 and anti-HPV 18 type specific neutralizing antibody level on day 0 (before the 1st dose) ,six month after the dose 1 (before the 3rd dose) and one month after dose 3

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, Ph. D., Study Chair — Xiamen University; Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China